CLINICAL TRIAL: NCT00616954
Title: An Investigator Initiated, Prospective, Randomized, Controlled Study in Order to Evaluate the Effect of Anti-thymocyte Globulin (Fresenius ATG) on Engraftment, Graft Versus Host Disease (GVHD) and Graft Versus Leukemia (GVL) Effect in Haplo-identical Allogeneic Hematopoietic Stem-cell Transplantation
Brief Title: A Study to Evaluate the Effect of ATG-F on Engraftment, Graft Versus Host Disease (GVHD) and Graft Versus Leukemia (GVL) Effect in Haplo-identical SCT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Hadassah Medical Organization, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYS-06-HMO-CTIL
Record Dates: First submitted 2008-01-22; First posted 2008-02-15 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2009-08

CONDITIONS: Allogeneic Haplo-Stem Cell Transplatation (SCT); Graft Versus Host Disease
Keywords: mismatched; Stem cell transplatation; Bone marrow transplantation; T cell depletion; engraftment; Patients undergoing allogeneic haplo-SCT
MeSH Terms: conditions — Graft vs Host Disease

ARMS (2):
- 1 (Experimental): with ATG-F
  Interventions: Drug: ATG-F
- 2 (No Intervention): control

INTERVENTIONS:
Drug: ATG-F — ATG-f
  Arms: 1

SUMMARY:
This study is planned to evaluated whether ATG is needed in haploidentical stem cell transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 3-70 years old with a disease necessitating allogeneic SCT.
2. Patients must have a mismatched donor willing and capable of donating peripheral blood stem cells and/or bone marrow progenitor cells using conventional techniques, and lymphocytes if indicated (mismatched defined as 3/6-4/6 HLA matching).
3. Each patient / patient's guardian must sign written informed consent.
4. Patients must have an ECOG PS ≤ 2; Creatinine <2.0 mg/dl; Ejection fraction >40%; DLCO >50% of predicted; Serum bilirubin <3 gm/dl; elevated GPT or GOT >3 x normal values.

Exclusion Criteria:

1. Not fulfilling any of the inclusion criteria.
2. Active life-threatening infection.
3. Overt untreated infection.
4. Known hypersensitivity to ATG.
5. HIV seropositivity, Hepatitis B or C antigen positivity with evidence of active hepatitis.
6. Pregnant or lactating women.
7. Donor contraindication (HIV seropositive confirmed by Western Blot Hepatitis B antigenemia; positive HCV antibodies with positive HCV PCR; evidence of bone marrow disease; unable to donate bone marrow or peripheral blood due to concurrent medical condition).
8. Inability to comply with study requirements.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Day of day of neutrophil engraftment (ANC>0.5x10^9/L) | 30 days
Day of platelet engraftment >25x10^9/L | 30 days

SECONDARY OUTCOMES:
AGVHD occurrence | 100 days
DFS at 100 days | 100 days
Day of platelet engraftment >50x10^9/L | 100 days
Time to AGVHD | 100 days
AGVHD grade | 100 days
OS | 100 days
Infections incidence | 100 days
TRM | 100 days
TRT | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y Shapira, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel